CLINICAL TRIAL: NCT06508567
Title: Salvage MR-guided High-Dose-Rate Brachytherapy for Prostate Bed Recurrence After Radiotherapy in the PSMA PET Scan Era
Acronym: SHAPE-PSMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-6023
Record Dates: First submitted 2024-03-15; First posted 2024-07-18 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer Recurrent; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2xHDR Brachytherapy (Experimental): Salvage MR-guided High-Dose-Rate Brachytherapy for Prostate Bed recurrence after Postoperative Radiotherapy.
  Interventions: Radiation: High Dose Rate Brachytherapy

INTERVENTIONS:
Radiation: High Dose Rate Brachytherapy — 2 fractions of MRI-guided HDR Brachytherapy (13Gy each) delivered over 14 days (± 7 days).

SUMMARY:
This is an interventional, single-centre, single-arm, non-randomized, prospective, feasibility trial investigating salvage MR-guided High-Dose-Rate brachytherapy for prostate bed recurrence after postoperative radiotherapy.

DETAILED DESCRIPTION:
Patients who received previous adjuvant or salvage radiotherapy to the prostate bed >

Isolated prostate bed recurrence based on PSMA PET, biopsy-proven, and MR visible >

Baseline: QoLs questionnaires, PSA, pelvic magnetic resonance imaging (MRI) scan for RT planning >

Two fractions of 13 Gy each delivered over 7-21 days. GTV(HDR) delineation (based on MRI-guided and PSMA PET, biopsy data as applicable) >

Follow-Up after treatment 60 months: PSA, CTCAE v5.0, MRI pelvis +/- PSMA-PET scan (optional at 24 months)

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received previous RT to the prostate bed +/- pelvic nodal regions
2. Prostate-bed recurrence identified by biopsy and/or MRI and/or PSMA-PET scan
3. At least two continuous PSA elevations post RT and PSA above 0.2 ng/dl
4. With or without ADT PSA doubling time from nadir greater than 6 months
5. ECOG 0-2
6. Age greater than 18 years

Exclusion Criteria:

1. Radiological (e.g. PSMA PET, CT, MRI or bone scan) evidence of or distant metastases
2. History of ≥G3 gastrointestinal (GI) and genitourinary (GU) toxicities following RT
3. Any contraindications to MR and/or brachytherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-08-08 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Dosimetry Parameters | 5 Years
  As this is a safety and feasibility study, the PTV coverage could be compromised to meet the OAR constraints
Acute toxicity assessed by CTCAE V5.0 (Grade ≥3) | 5 Years
  Determine the number of patients with late genitourinary, gastrointestinal and/or sexual toxicities as a result of salvage HDR Brachytherapy treatment at a grade ≥3

SECONDARY OUTCOMES:
Biochemical Control assessed by PSA | 5 Years
  Determine the number of patients demonstrating biochemical control of PSA following salvage HDR Brachytherapy treatment.
Local Disease Control | 2 Years
  Assessed by MRI/PSMA-PET imaging at 2 years
Changes in Quality of Life | 5 years
  Assessed with EPIC Quality of Life scores yearly for 5 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada